CLINICAL TRIAL: NCT04554056
Title: A Phase II/III,Multi-Center,Randomized,Double-blind,Active-Controlled Trial to Compare the Efficacy , Safety and Immunogenicity of MW05 and PEG-rhG-CSF in Prophylactic Treatment for Chemotherapy-Induced Neutropenia
Brief Title: Trial to Compare the Efficacy and Safety Of MW05 and PEG-rhG-CSF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MW05-2020-CP301
Record Dates: First submitted 2020-07-27; First posted 2020-09-18 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MW05 300μg/kg (Experimental): Subjects will receive MW05(300 μg/kg s.c.) on day 3 of each cycle (6~10 a.m.)
  Interventions: Drug: MW05
- MW05 500μg/kg (Experimental): Subjects will receive MW05(500 μg/kg s.c.) on day 3 of each cycle (6~10 a.m.)
  Interventions: Drug: MW05
- PEG-rhG-CSF (Active Comparator): Subjects will receive PEG-rhG-CSF(100 μg/kg s.c.) on day 3 of each cycle (6~10 a.m.)
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: MW05 — Recombinant (yeast secreted) human serum albumin-human granulocyte colony stimulating factor (I) fusion protein injection
  Other Names: MW05 injection
  Arms: MW05 300μg/kg; MW05 500μg/kg
Drug: PEG-rhG-CSF — PEGylated Recombinant Human Granulocyte Colony-Stimulating Factor
  Other Names: PEG-rhG-CSF injection
  Arms: PEG-rhG-CSF

SUMMARY:
In the study, subjects will scheduled to undergo four 21-days cycles of chemotherapy treatment. Three group were treated with MW05 300 μg/kg or MW05 500 μg/kg or PEG-rhG-CSF 100 μg/kg on the 3th day of each cycle randomized 1:1:1 .

The dose of the experimental drug MW05 in phase III were determined by independent data monitoring committee (IDMC) according to the efficacy and safety of phase II. Subjects were randomly divided into two groups 1:1 to received either MW05 or PEG-rhG-CSF(100 μg/kg) on the 3th day of each chemotherapy cycle.

DETAILED DESCRIPTION:
Study Stage: Phase II/III Study Population Female patients with breast cancer will be enrolled to receive at least 4 cycles of TC chemotherapy, that is: Docetaxel 75 mg/m2 and Cyclophosphamide 600 mg/m2.

Study Design: A multi-center, randomized, open-label, active-controlled phase II/III clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. 18～70 years old female(including threshold)
2. Diagnosed with breast cancer .
3. Weight≥45kg.
4. Patients planned to receive TC chemotherapy.
5. ECOG ≤ 1
6. Estimated survival time ≥ 3 months, and could received at least 4 cycles chemotherapy treatment.
7. Have suitable organs and hematopoietic function
8. ECG examination is normal or abnormal has no clinical significance.
9. B-ultrasound examination of abdomen showed no obvious abnormality of spleen.
10. Willing to sign the informed consent form and able to comply with protocol requirements.
11. Non-menopausal or non-surgically sterilized female subjects, the blood pregnancy test results must be negative at the time of screening, and within at least 3 months from the signing of the informed consent form to the end of the last administration, consent to abstinence or the use of effective contraceptive methods.

    -

Exclusion Criteria:

1. History of other malignant tumors (skin basal cell carcinoma, skin squamous cell carcinoma and / or carcinoma in situ after radical resection can be included in the group after being cured for more than 5 years)
2. Primary hematological diseases, including but not limited to myelodysplastic syndrome, aplastic anemia, sickle cell anemia and other hematological diseases that affect bone marrow hematopoiesis.
3. With known central nervous system metastasis or suspected central nervous system metastasis based on clinical manifestations.
4. With previous history of bone marrow transplantation and / or stem cell transplantation.
5. Currently uncontrolled infections or have received systematic anti-infective therapy within 72 hours before randomization.
6. Serious chronic diseases of important organs such as kidney and liver.
7. Severe heart disease, including but not limited to:history of congestive heart failure (New York College of Cardiology [NYHA] II or higher heart disease)Angina pectoris that needs to be treated with anti-angina pectoris drugsUncontrollable hypertension (systolic blood pressure ≥ 180 mmHg and / or diastolic blood pressure ≥ 100 mmHg)Arrhythmias requiring drug treatment
8. Severe diabetes (such as fundus disease or diabetic foot), or blood sugar is still not well controlled after active treatment.
9. Surgery within 2 weeks before chemotherapy or radiotherapy within 4 weeks (except for patients whose physical condition has recovered and can accept the relevant procedures of this study, as determined by the researchers)
10. Adverse reactions from previous treatments failed to recover to CTCAE v5.0 score ≤ 1 (except for alopecia and other toxic reactions that researchers believe do not affect the safety of this chemotherapy)
11. According to the researchers, there are serious risks to the safety of patients or concomitant diseases that affect the completion of the study.
12. Participated in clinical trials of any other drugs within 4 weeks.
13. Received the same efficacy drugs(such as PEG-rhG-CSF or rhG-CSF, etc.) are still in 5 half-lives or within 28 days (whichever is shorter).
14. With allergic disease or allergic constitution, and who have previously been allergic to any drug or its components in this trial.
15. Active hepatitis B (HBsAg positive and HBV-DNA copy number greater than the normal limit) and / or active hepatitis C (hepatitis C virus antibody positive and HCV-RNA copy number greater than the normal limit) and / or human immunodeficiency virus antibody positive and / or Treponema pallidum antibody.
16. Drug abuse. history or drug abusers
17. Pregnant or lactating women
18. Who have been judged by the researchers to be unsuitable for selection or who are not suitable for other reasons

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with breast cancer who require chemotherapy and are planned to receive at least 4 cycles of TC chemotherapy, namely Docetaxel 75 mg/m2 and Cyclophosphamide 600 mg/m2
Enrollment: 586 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study will be to evaluate the efficacy of MW05 pre-filled syringe as compared to PEG-rhG-CSF standard dosing (6 mg) in the first chemotherapy cycle. | in cycle 1（each cycle is 21 days）
  The primary endpoint will be the duration of grade 4 (severe) neutropenia - the number of days in which the patient has had an absolute neutrophil count (ANC <0.5 x 109/L) observed in chemotherapy cycle 1.

SECONDARY OUTCOMES:
The duration of grade 4 neutropenia in cycle 2~4 assessed by ANC（ANC < 0.5 × 109/L） | in cycles 2-4, in overall 3 cycles（each cycle is 21 days）
  The duration of grade 4 neutropenia (ANC< 0.5 × 109/L)
The incidence of grade 4 neutropenia in cycle 1~4 assessed by ANC（ANC < 0.5 × 109/L） | through study completion, in overall 4 cycles（each cycle is 21 days）
  The incidence rate of grade 4 neutropenia (ANC< 0.5 × 109/L)
The incidence of grade 3 or 4 neutropenia in cycle 1~4 assessed by ANC（ANC < 1.0 × 109/L and ANC < 0.5 × 109/L, respectively） | through study completion, in overall 4 cycles（each cycle is 21 days）
  The incidence rate of grade 3 or 4 neutropenia (ANC < 1.0 × 109/L and ANC< 0.5 × 109/L, respectively)
The duration of grade 3 or 4 neutropenia In cycle 1~4 assessed by ANC（ANC < 1.0 × 109/L and ANC < 0.5 × 109/L, respectively） | through study completion, in overall 4 cycles（each cycle is 21 days）
  The duration of grade 3 or 4 neutropenia (ANC < 1.0 × 109/L and ANC< 0.5 × 109/L, respectively)
Incidence of febrile neutropenia (FN) (defined as ANC < 1.0×109/L; a single measurement of body temperature > 38.3°C or a temperature ≥ 38.0 °C sustained over 1 h) | through study completion, in overall 4 cycles（each cycle is 21 days）
  Rate of febrile neutropenia (FN) (defined as ANC < 1.0×109/L; a single measurement of body temperature > 38.3 °C or a temperature ≥ 38.0 °C sustained over 1 h)
The proportion of subjects rescued by short-acting G-CSF in cycle 1~4. | through study completion, in overall 4 cycles（each cycle is 21 days）
  The proportion of received short-acting G-CSF.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Affiliated Cancer Hospital, Shanghai, China